CLINICAL TRIAL: NCT00051246
Title: Relational Group Intervention for Postpartum Depression
Brief Title: Group Therapy for Postpartum Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH062054 (NIH); R01MH062054 (NIH)
Record Dates: First submitted 2003-01-07; First posted 2003-01-08 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Depression, Postpartum
MeSH Terms: conditions — Depression, Postpartum | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 M-ITG (Active Comparator): Mother-infant group psychotherapy
  Interventions: Behavioral: Mother-Infant Group Psychotherapy
- 2 - IPT (Active Comparator): Individual interpersonal psychotherapy
  Interventions: Behavioral: Interpersonal Psychotherapy

INTERVENTIONS:
Behavioral: Mother-Infant Group Psychotherapy — Mother-infant group psychotherapy consists of weekly 2.5-hour psychotherapy sessions comprised of mother's group therapy, infant developmental therapy, and mother-infant dyadic psychotherapy. Group treatment will last 15 weeks.
  Arms: 1 M-ITG
Behavioral: Interpersonal Psychotherapy — Individual psychotherapy treatment focuses on role transition, interpersonal relationships, and loss. Individual treatment period will last 15 weeks.
  Arms: 2 - IPT

SUMMARY:
This study will compare standard individual treatment to group therapy for the treatment of postpartum depression.

DETAILED DESCRIPTION:
Ten to twenty percent of new mothers experience major depression in the postpartum period or postpartum depression (PPD). This condition poses a risk for disturbances in the mother-infant relationship as well as for developmental delays and subsequent psychopathology in their children. Thus, and investigation of the efficacy of a relational approach that focuses on improving the mother's sense of competence in the parenting role, and reducing depressive symptoms and social isolation through group therapy is warranted.

Patients are randomly assigned to either relational group treatment or to standard individual treatment. Assessments of maternal and infant functioning, mother-infant and father-infant relations, parenting stress, and marital conflict and conducted pre- and post-treatment, at 12 months post-treatment, and when infants are 12 and 24 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Major depression with an infant under 7 months of age

Exclusion Criteria:

* Bipolar disorder
* Schizophrenia
* Organic brain syndrome
* Antisocial personality disorder
* Current psychosis or mania
* Lifetime history of mental retardation
* Current alcohol or substance abuse
* Cognitive disability
* Infants born more than 6 weeks premature or with major medical conditions or developmental disabilities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2002-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Reduction of depression as measured by the Hamilton Rating Scale for Depression (HRSD) | Measured at post-treatment and Month 12 follow-up

SECONDARY OUTCOMES:
Improvement in parent-infant interactions as measured by the Early Relational Assessment (ERA) | Measured at post-treatment, Month 12 follow-up, and 12 and 24 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Roseanne Clark, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Dept. of Psychiatry, Madison, Wisconsin, United States